CLINICAL TRIAL: NCT01146236
Title: Sutures vs Staples for Wound Closure in Orthopaedic Surgery: A Randomized Controlled Trial
Brief Title: Sutures Versus Staples for Wound Closure in Orthopaedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other); Gibson Orthopaedic Fund for Research and Education (Other)
Responsible Party: Principal Investigator, Dr. Jesse Shantz, Orthopedic Surgeon, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WCRCT
Record Dates: First submitted 2010-06-14; First posted 2010-06-17 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Surgical Wound Infection
Keywords: Surgical; Infection; Post-operative; Sutures; Staples
MeSH Terms: conditions — Surgical Wound Infection; Infections | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sutures (Active Comparator): Orthopedic surgical wound closed with sutures
  Interventions: Device: Sutures
- Staples (Active Comparator): Orthopedic surgical wound closed with metallic staples
  Interventions: Device: Staples

INTERVENTIONS:
Device: Sutures — Orthopedic surgical wounds closed with sutures
  Arms: Sutures
Device: Staples — Orthopedic surgical wounds closed with metallic staples
  Arms: Staples

SUMMARY:
The trial is a randomized, controlled trial. Adult patients undergoing orthopaedic surgical procedures would be randomized to one of two groups for surgical wound closure, skin sutures or skin staples. The primary outcome measures would be surgical site infection indicated by the use of oral or intravenous antibiotics for suspected wound infection and/or re-operation at the same site. Patients would be followed up as per their usual post-operative course for a total of three months in the trauma and spine population and six months in the total joint arthroplasty population. It is hypothesized that wounds closed with sutures and staples will have similar infection rates as defined by the use of antibiotics or reoperation.

DETAILED DESCRIPTION:
To date, there is no clear consensus on the method that is best for closure of surgical wounds in orthopaedic surgery. Orthopaedic surgeons have a multitude of wound closure habits. A recent meta-analysis comparing staples to sutures in wound closure demonstrated a three-fold increase in infection in stapled wounds compared to sutured wounds. The studies used in the meta-analysis were primarily of poor methodological quality.

A large, well-designed randomized, controlled trial is needed to guide orthopedic surgeons in their choice of wound closure materials. This study would attempt to provide information on the use of sutures versus skin staples and the effect on the development of surgical site infections in adults undergoing orthopaedic procedures.

A parallel group randomized controlled trial with institutional review board approval will be conducted. Patients will be randomized intraoperatively to have skin wounds closed with sutures or staples. Dressings will be used to maintain blinding of participants and outcome assessors. The primary outcome measure will be infections adjudicated by a blinded data safety monitoring committee. Suspected infections will be defined by: Use of antibiotics or reoperation for infection at the operative site within three months (six months for arthroplasty subgroup) The independent review, board blinded to treatment assignment, will adjudicate suspected infections based on clinical data. A cost analysis will also be performed to compare the costs associated with wounds closed with sutures and staples from a health care institution perspective.

All data will be analyzed by a blinded epidemiologist. Dichotomous primary and secondary outcome measures will be analyzed using the Chi-squared statistic. Continuous outcome measures will be analyzed using Student's t-test. Subgroup analysis will compare infection rates using sutures versus staples in each anatomic area (upper extremity, pelvis/acetabulum, hip/femur, knee, ankle). A further subgroup analysis will be conducted comparing trauma patients to elective patients. Non-infected revision surgery will also be compared to primary surgery.

It is hypothesized that wounds closed with sutures and staples will have similar infection rates as defined by the use of antibiotics or reoperation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* All open orthopedic procedures
* Largest wound >2cm in length

Exclusion Criteria:

* Open fracture
* Known nickel allergy
* Active infection (any site)
* Chemotherapy during study period (1 month prior until end of follow-up)
* Radiation therapy to surgical site (1 month prior until end of follow-up)
* Foot surgery (any site)
* Hand surgery (including carpal surgery)
* Arthroscopic procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2010-07; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 6 months
  Suspected cases will be identified by one or all of the following: use of intravenous antibiotics, use of oral antibiotics (patient self-reported), re-operation at same site. A blinded committee will adjudicate each suspected case and determine true infections using available clinical information. Agreement will be determined by vote.

SECONDARY OUTCOMES:
Additional healthcare contact related to their surgery | 6 months
  As defined by self-reported visits to other healthcare professionals.
Dressing changes by homecare/patient at home | 6 months
  Defined by homecare consult records and patient self-report
Length of stay | 6 months
  Based on admission and discharge dates
Wound drainage | 6 months
  As defined by necessity for dressing changes after 72 hours for fluid leakage
Wound necrosis | 6 months
  Evidence of marginal skin death at the surgical site as evidenced by skin slough, blackening or liquefaction
Patient satisfaction with wound appearance | 6 months
  Using visual analogue scale
Visual analogue pain score for suture/staple removal | 2 weeks post-operative
  Patients will rate the pain experienced in removing the wound closure materials in clinic prior to unblinding.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Shantz, MD, MBA, Principal Investigator — University of Manitoba
Locations (3):
- Canada (3):
  - Concordia Hip and Knee Institute, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba
  - Pan Am Clinic, Winnipeg, Manitoba

REFERENCES:
- [Derived] Slade Shantz JA, Vernon J, Morshed S, Leiter J, Stranges G. Sutures versus staples for wound closure in orthopaedic surgery: a pilot randomized controlled trial. Patient Saf Surg. 2013 Feb 9;7(1):6. doi: 10.1186/1754-9493-7-6. PMID 23394586
- [Derived] Shantz JA, Vernon J, Leiter J, Morshed S, Stranges G. Sutures versus staples for wound closure in orthopaedic surgery: a randomized controlled trial. BMC Musculoskelet Disord. 2012 Jun 6;13:89. doi: 10.1186/1471-2474-13-89. PMID 22672186